CLINICAL TRIAL: NCT03614936
Title: Study of a Simplified Geriatric Evaluation Performed by Oncologists Prior to Cancer Treatment by Radiotherapy or Chemotherapy in Subjects Aged 70 Years or Older With Inoperable Squamous Cell Cancer of the Head and Neck
Acronym: ELAN-ONCOVAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-A00888-35; 2013/1962 (Other: CSET number)
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Inoperable Squamous Cell Cancer of the Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inoperable squamous cell cancer of the head and neck: patients 70 years of age or older with ENT carcinoma
  Interventions: Other: Geriatric Screening Test G8; Other: Geriatric fragility test GERICO

INTERVENTIONS:
Other: Geriatric Screening Test G8 — Geriatric screening test (Oncodage-G8). The oncologist realizes it and proposes the oncological treatment which seems to him then the most adapted (treatment which can be different from that proposed after the oncological evaluation only).
Other: Geriatric fragility test GERICO — GERICO geriatric frailty test (if possible the same day as the G8 and in any case in the same week): Realized by the oncologist, it includes:
  * the socio-cultural evaluation scale,
  * the ADL autonomy questionnaire,
  * assessment of locomotor disorders,
  * nutritional assessment,
  * the MMSE Cognitive Function Evaluation Questionnaire,
  * the GDS-4 mood rating scale,
  * the comorbidity assessment test (Charlson Index)

SUMMARY:
Use by Oncologists of Validated Geriatric Assessment Tools: G8 Screening Test and Certain Tests for Thorough Geriatric Evaluation

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 70 or over
* Carrier of squamous cell carcinoma of the head and neck, locally advanced undergoing treatment by radiotherapy or metastatic / recurrence not accessible to treatment curative locoregional under treatment with chemotherapy.
* Patient likely to be eligible for ELAN-RT or ELAN-FIT or ELAN-UNFIT trials.
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Person deprived of liberty or under guardianship,
* Presence of a neuro-psychological condition, family, social, or geographical, which may hinder the smooth running of the study.
* Patient expressing opposition to participation in this study

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients 70 years of age or older with ENT carcinoma
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-06-11 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Completion rate | Up to 1 year
  Rate of completion of each of the geriatric fragility test questionnaires and the G8 questionnaire and duration of the geriatric evaluation performed by the oncologist

CONTACTS AND LOCATIONS:
Overall Officials: Joel GUIGAY, MD, PhD, Study Chair — Centre Antoine Lacassagne
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided